CLINICAL TRIAL: NCT03555851
Title: Elucidation of Factors Predicting Efficacy and Toxicity of Post Transplantation Cyclophosphamide (PTCy) as a Strategy for Graft Versus Host Disease Prevention in Haploidentical, Matched Related Donor and Matched Unrelated Donor Peripheral Blood Hematopoietic Cell Transplantation
Brief Title: Factors Affecting Post-transplant Cyclophosphamide (PTCy) Efficacy
Status: Recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00081375; LCI-HEM-HCT-PTCY-001 (Other: Atrium Health); Pro00024582 (Other: Advarra IRB); NCI-2024-06503 (Other: National Cancer Institute)
Record Dates: First submitted 2018-05-02; First posted 2018-06-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Leukemia, Not Otherwise Specified; Leukemia, Other
MeSH Terms: conditions — Leukemia | interventions — Cyclophosphamide; Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal swabs, whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recipient: Cyclophosphamide
  Interventions: Drug: Cyclophosphamide; Other: Specimen collection
- Donor: Specimen collection
  Interventions: Other: Specimen collection

INTERVENTIONS:
Drug: Cyclophosphamide — Pharmacogenomics of candidate genes and pharmacokinetic analyses of cyclophosphamide administered as part of a reduced intensity conditioning (RIC) regimen and as post-transplant GVHD prophylaxis will be examined.
  Groups: Recipient
Other: Specimen collection — Buccal swabs will be obtained from donors for pharmacogenomics.

SUMMARY:
This study will examine the influence of donor and recipient pharmacogenetics (PG), drug pharmacokinetics (PK), and T cell phenotypes and how it may permit a tailored dosing strategy to improve the therapeutic index of post-transplant cyclophosphamide (PTCy) and optimize the graft versus tumor effect, while minimizing acute and chronic graft versus host disease (GVHD).

DETAILED DESCRIPTION:
The primary objective of this single-arm, pilot study is to determine whether pharmacogenetics (PG) of Cy-related candidate genes from the recipients and/or donors (haploidentical and matched related donor HCTs only) germ-line DNA is associated with incidence and severity of acute and chronic GVHD. Secondary objectives include determining whether pharmacogenetics (PG) of Cy-related candidate genes from the recipients and/or donors (haploidentical and matched related donor HCTs only) germ-line DNA is associated with Cy (and metabolites) exposure and toxicities; quantifying Cy (and related metabolites) exposure measured as the area under the concentration time curve (AUC) from zero to 24 hours both before (day -6) and after transplant (day +3), and correlate exposure with incidence of acute and chronic GVHD, and Adverse Events of Special Interest (AESIs); and determining whether immune activation or polarization prior to or following Cy GVHD prophylaxis is associated with grade of acute or chronic GVHD grade and AESIs. Safety objects include evaluating Cy administered, adverse events of special interest (including deaths while on study therapy), selected laboratory parameters (including time to neutrophil recovery), and immunosuppressant concomitant medications administration. Initially, 20 participants (HCT recipients and their respective haploidentical or matched related donors) will be enrolled with a subsequent 100 additional subjects enrolled.

ELIGIBILITY:
Inclusion Criteria

Recipients and donors must meet all of the following applicable inclusion criteria to participate in this study:

1. Informed consent and HIPAA authorization for release of personal health information signed by the subject.
2. Age ≥ 18 years at the time of consent.
3. Subject is scheduled as a recipient or respective donor (Donor consent/participation is not required for subjects undergoing matched unrelated donor HCT) for the following hematopoietic stem cell transplants (HCT) procedures using a non-myeloablative regimen at Levine Cancer Institute (LCI), and has been deemed a qualified candidate by his/her physician, per LCI medical standards: haplo-identical donor HCT, match related donor (MRD) HCT, matched unrelated donor (MUD) HCT.
4. Recipient only: Planned post-transplant cyclophosphamide
5. As determined by the enrolling physician, ability of the subject to understand and comply with study procedures for the entire length of the study

Exclusion Criteria

Subjects meeting any of the criteria below may not participate in the study:

1. Recipient only (applies only to haplo-identical and MRD HCT recipients; not required for MUD HCT recipients): Does not have a respective donor who is willing to sign informed consent for participation in this study.
2. Recipient only: Treatment with any investigational drug within 30 days prior to day -6 of treatment
3. Donor only (applies only to haplo-identical and MRD HCTs; donor participation is not required for MUD HCTs): Does not have a respective recipient who is willing to sign informed consent for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are scheduled as a recipient or respective donor for the following hematopoietic stem cell transplants (HCT): haplo-identical donor HCT, match related donor (MRD) HCT, matched unrelated donor (MUD) HCT.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-07-13 (Actual); Primary Completion 2033-10 (Estimated); Study Completion 2035-08 (Estimated)

PRIMARY OUTCOMES:
Comparison of Cy cMax Values | Approx. 24 mos
  Evaluation and comparison of average Day 3 Cy cMax values between subjects who experience acute GVHD versus subjects who do not experience acute GVHD

SECONDARY OUTCOMES:
Incidence of chronic GVHD | Approx. 24 mos
  Calculated for each subject as a binary variable indicating whether or not subject experienced chronic GVHD
Cy exposure | Approx. 10 days
  Cy (and related metabolites) exposure will be calculated using area under the concentration curve (AUC). This will be accomplished using the trapezoidal approximation, and will be calculated over the 24 hour period following first pre-transplant dose of Cy and over the 24 hour period following post-transplant dose of Cy.
Toxicities | Approx. 180 days
  The incidence of adverse events of special interests will be collected according to CTCAE version 4.03
Pharmacogenetics of Cy-related genes | Approx. 24 mos
  Evaluation of the prognostic value of pharmacogenetics (PG) of Cy-related candidate genes from the recipient's germ-line DNA, using logistic regression, on the incidence and severity of acute and chronic GVHD. PG of Cy-related candidate genes will be performed on 12 genes. Genes encoding CYP enzymes will be classified into metabolizer status and other genes will be classified as either wild type, heterozygous, or homozygous variants.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksander Chojecki, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No